CLINICAL TRIAL: NCT04785599
Title: Effectiveness of Lymphedema Prevention Programs After Lymph Node Emptying in Breast Cancer: A Randomized Clinical Trial
Brief Title: Lymphedema Prevention After Lymph Node Emptying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIBSP-EPC-2011-87
Record Dates: First submitted 2021-01-26; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Lymphedema; Breast Cancer; Prevention; Rehabilitation
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group EC1: Exercices, informative talk (Experimental): Group EC1 carried out the conventional prevention program consisting of an informative talk and an exercise program
  Interventions: Behavioral: Exercices; Behavioral: Informative talk
- Group ECCP2: Exercices, informative talk, compression garment (Experimental): Group ECCP2 carried out the same program but with the addition of a prophylactic compression garment
  Interventions: Behavioral: Exercices; Behavioral: Informative talk; Device: Compression garment

INTERVENTIONS:
Behavioral: Exercices — An exercise program. Seven days after lymph node removal, participants began this program at the physiotherapy department. They attended two weekly sessions of 60 minutes each. The sessions at the centre continued for 12 weeks. The program consisted of aerobic exercise, in combination with resistance and stretching exercises.
Behavioral: Informative talk — An informative talk: Patients attended a one-hour long talk about lymphedema. The topics covered were a description of the condition, the risks, and preventive measures to include in their daily life. The recommended measures were those from the general consensus of the International Lymphedema Society, the Spanish Rehabilitation Society and The National Breast and Ovarian Cancer Center
Device: Compression garment — Wearing a flat knit compression garment (CG), class 1. Participants were recommended to wear this CG for an average of 8 hours during the daytime for the first 3 months after surgery, and to remove it at night.
  From the fourth month onwards, use of the garment was reduced to 2 hours a day, coinciding with exercises and physical activity.
  Arms: Group ECCP2: Exercices, informative talk, compression garment

SUMMARY:
ABSTRACT Object: The impact of morbidity and the deterioration in health-related quality of life for patients with lymphedema after axillary lymph node dissection for breast cancer justify the implementation of prevention programs to decrease the incidence of this chronic condition. The aim was to compare the effectiveness of an experimental prevention program with that of our conventional prevention program.

Methods: Clinical randomized trial in two parallel groups over a two-year period.

Key words: lymphedema, breast cancer, prevention, rehabilitation

DETAILED DESCRIPTION:
This was a single-centre, open-label, controlled, randomized clinical trial. Patients were recruited from the Breast Pathology Unit at Hospital de la Santa Creu i Sant Pau (HSCSP), a tertiary referral hospital in Barcelona between March 2011 and April 2013. The inclusion criteria were as follows:

* Patients between 18 and 85 years
* Having undergone a lymph node dissection as part of treatment for primary breast neoplasm
* Acceptance of the study conditions and signing of the informed consent

Exclusion criteria were:

* tumour recurrences
* metastatic cancer
* open wounds or loss of skin integrity
* dependency or deterioration of higher functions
* arterial insufficiency and deep vein thrombosis
* acute heart failure
* severe peripheral neuropathy
* lymphedema Patients included in the study were randomized to one of two groups. Group 1(G1) carried out the conventional prevention program consisting of an informative talk and an exercise program. Group 2(G2) carried out the same program but with the addition of a prophylactic compression garment.

The program common to both groups consisted of:

1. An informative talk: Patients attended a one-hour long talk about lymphedema. The topics covered were a description of the condition, the risks, and preventive measures to include in their daily life. The recommended measures were those from the general consensus of the International Lymphedema Society, the Spanish Rehabilitation Society and The National Breast and Ovarian Cancer Center (J.González-Sánchez y Sánchez- Mata F 2010) (See tables 1 and 2).
2. An exercise program. Seven days after lymph node removal, participants began this program at the physiotherapy department. They attended two weekly sessions of 60 minutes each. The sessions at the centre continued for 12 weeks. The program consisted of aerobic exercise, in combination with resistance and stretching exercises.

Group 2 (experimental) was also prescribed:

• A flat knit compression garment (CG), class 1. Participants were recommended to wear this CG for an average of 8 hours during the daytime for the first 3 months after surgery, and to remove it at night. From the fourth month onwards, use of the garment was reduced to 2 hours a day, coinciding with exercises and physical activity.

The study was evaluated and authorized by the Ethics Committee at Hospital de la Santa Creu i Sant Pau (HSCSP), code IIBS-EPC-2011-87. All patients signed the written informed consent form.

Evaluations All patients were evaluated at the start of the study, at the end of the exercise prevention program, at 6 months, and at one and two years.

In all the evaluations, we measured the volume of the upper extremities following the lymphedema calculation formula based on the truncated cone, validated and published by the Spanish Society of Physical Medicine and Rehabilitation (SERMEF).

Lymphedema was defined as a difference of more than 200 ml in volume between the upper extremities, or as a difference of 10% in volume between the two upper limbs (SERMEF 2012).

We recorded all the parameters of the history and general clinical examination, TNM stage, performed treatments, number of resected nodes and complications. Compliance with all the components of each program was monitored. Data regarding presence at the talk and at the exercise program sessions at the centre were recorded by calendar. Home compliance was monitored through personal interviews at 6 months, 1 year and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone a lymph node dissection as part of treatment for primary breast neoplasm
* Acceptance of the study conditions and signing of the informed consent

Exclusion Criteria:

* Tumour recurrences
* Metastatic cancer
* Open wounds or loss of skin integrity
* Dependency or deterioration of higher functions
* Arterial insufficiency and deep vein thrombosis
* Acute heart failure
* Severe peripheral neuropathy
* Lymphedema

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-10-03 (Actual); Primary Completion 2011-10-03 (Actual); Study Completion 2015-04-13 (Actual)

PRIMARY OUTCOMES:
Measure of arms volume | All patients were evaluated at the start of the study
  Lymphedema was defined as a difference of more than 200 ml in volume between the upper extremities, or as a difference of 10% in volume between the two upper limbs (SERMEF 2012).
Measure of arms volume | All patients were evaluated at 3 months from beginning
  Lymphedema was defined as a difference of more than 200 ml in volume between the upper extremities, or as a difference of 10% in volume between the two upper limbs

OTHER OUTCOMES:
Measure of arms volume | All patients were evaluated at 6 months from beginning
  Lymphedema was defined as a difference of more than 200 ml in volume between the upper extremities, or as a difference of 10% in volume between the two upper limbs
Measure of arms volume | All patients were evaluated at 12 months from beginning
  Lymphedema was defined as a difference of more than 200 ml in volume between the upper extremities, or as a difference of 10% in volume between the two upper limbs
Measure of arms volume | All patients were evaluated at 24 months from beginning
  Lymphedema was defined as a difference of more than 200 ml in volume between the upper extremities, or as a difference of 10% in volume between the two upper limbs

CONTACTS AND LOCATIONS:
Overall Officials: Maria José Nadal Castells, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau

IPD SHARING:
Plan to Share IPD: Yes
We recorded all the parameters of the history and general clinical examination, TNM stage, performed treatments, number of resected nodes and complications. Compliance with all the components of each program was monitored. Data regarding presence at the talk and at the exercise program sessions at the centre were recorded by calendar. Home compliance was monitored through personal interviews at 6 months, 1 year and 2 years.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Supporting information is already available
Access Criteria: Free access
URL: https://www.educacion.gob.es/teseo/irGestionarConsulta.do

REFERENCES:
- [Background] Baumann FT, Reike A, Hallek M, Wiskemann J, Reimer V. Does Exercise Have a Preventive Effect on Secondary Lymphedema in Breast Cancer Patients Following Local Treatment? - A Systematic Review. Breast Care (Basel). 2018 Oct;13(5):380-385. doi: 10.1159/000487428. Epub 2018 May 3. PMID 30498426
- [Background] Boccardo FM, Ansaldi F, Bellini C, Accogli S, Taddei G, Murdaca G, Campisi CC, Villa G, Icardi G, Durando P, Puppo F, Campisi C. Prospective evaluation of a prevention protocol for lymphedema following surgery for breast cancer. Lymphology. 2009 Mar;42(1):1-9. PMID 19499762
- [Background] Cavanaugh KM. Effects of early exercise on the development of lymphedema in patients with breast cancer treated with axillary lymph node dissection. J Oncol Pract. 2011 Mar;7(2):89-93. doi: 10.1200/JOP.2010.000136. PMID 21731515
- [Background] Castro-Sanchez AM, Moreno-Lorenzo C, Mataran-Penarrocha GA, Aguilar-Ferrandiz ME, Almagro-Cespedes I, Anaya-Ojeda J. [Preventing lymphoedema after breast cancer surgery by elastic restraint orthotic and manual lymphatic drainage: a randomized clinical trial]. Med Clin (Barc). 2011 Jul 23;137(5):204-7. doi: 10.1016/j.medcli.2010.09.020. Epub 2010 Dec 8. Spanish. PMID 21145085
- [Background] Cheema BS, Kilbreath SL, Fahey PP, Delaney GP, Atlantis E. Safety and efficacy of progressive resistance training in breast cancer: a systematic review and meta-analysis. Breast Cancer Res Treat. 2014 Nov;148(2):249-68. doi: 10.1007/s10549-014-3162-9. Epub 2014 Oct 17. PMID 25324019
- [Background] De Miguel, C., Alonso, B., Hernandez, M., Crespo, M.P., Gil, M.S., 2010. Treatment with compression garments. Rehabilitation, 44 (51), 58-62.
- [Background] DiSipio T, Rye S, Newman B, Hayes S. Incidence of unilateral arm lymphoedema after breast cancer: a systematic review and meta-analysis. Lancet Oncol. 2013 May;14(6):500-15. doi: 10.1016/S1470-2045(13)70076-7. Epub 2013 Mar 27. PMID 23540561
- [Background] Gonzalez-Sanchez, J., and Sánchez- Mata, F., 2010. Quality of life, rating scales and preventive measures in lymphedema. Rehabilitation 44 (S1), 44-48.
- [Background] Hayes SC, Reul-Hirche H, Turner J. Exercise and secondary lymphedema: safety, potential benefits, and research issues. Med Sci Sports Exerc. 2009 Mar;41(3):483-9. doi: 10.1249/MSS.0b013e31818b98fb. PMID 19204604
- [Background] Kwan ML, Cohn JC, Armer JM, Stewart BR, Cormier JN. Exercise in patients with lymphedema: a systematic review of the contemporary literature. J Cancer Surviv. 2011 Dec;5(4):320-36. doi: 10.1007/s11764-011-0203-9. Epub 2011 Oct 16. PMID 22002586
- [Background] Kwan ML, Darbinian J, Schmitz KH, Citron R, Partee P, Kutner SE, Kushi LH. Risk factors for lymphedema in a prospective breast cancer survivorship study: the Pathways Study. Arch Surg. 2010 Nov;145(11):1055-63. doi: 10.1001/archsurg.2010.231. PMID 21079093
- [Background] Ochalek K, Partsch H, Gradalski T, Szygula Z. Do Compression Sleeves Reduce the Incidence of Arm Lymphedema and Improve Quality of Life? Two-Year Results from a Prospective Randomized Trial in Breast Cancer Survivors. Lymphat Res Biol. 2019 Feb;17(1):70-77. doi: 10.1089/lrb.2018.0006. Epub 2018 Oct 19. PMID 30339481
- [Background] Sagen A, Karesen R, Risberg MA. Physical activity for the affected limb and arm lymphedema after breast cancer surgery. A prospective, randomized controlled trial with two years follow-up. Acta Oncol. 2009;48(8):1102-10. doi: 10.3109/02841860903061683. PMID 19863217
- [Background] Sander, A.P., 2008. A safe and effective upper extremity resistive exercise program for woman post breast cancer treatment. Rehabilitation Oncology. 26(3), 3-10
- [Background] SERMEF. 2012. Applications. Lymphedema calculator for upper limb (Consulted on January 10, 2012). Available at: http://www.sermef.es/index.php.
- [Background] Singh B, Disipio T, Peake J, Hayes SC. Systematic Review and Meta-Analysis of the Effects of Exercise for Those With Cancer-Related Lymphedema. Arch Phys Med Rehabil. 2016 Feb;97(2):302-315.e13. doi: 10.1016/j.apmr.2015.09.012. Epub 2015 Oct 9. PMID 26440777
- [Background] Stout NL, Binkley JM, Schmitz KH, Andrews K, Hayes SC, Campbell KL, McNeely ML, Soballe PW, Berger AM, Cheville AL, Fabian C, Gerber LH, Harris SR, Johansson K, Pusic AL, Prosnitz RG, Smith RA. A prospective surveillance model for rehabilitation for women with breast cancer. Cancer. 2012 Apr 15;118(8 Suppl):2191-200. doi: 10.1002/cncr.27476. PMID 22488693
- [Background] Stout Gergich NL, Pfalzer LA, McGarvey C, Springer B, Gerber LH, Soballe P. Preoperative assessment enables the early diagnosis and successful treatment of lymphedema. Cancer. 2008 Jun 15;112(12):2809-19. doi: 10.1002/cncr.23494. PMID 18428212
- [Background] Temur K, Kapucu S. The effectiveness of lymphedema self-management in the prevention of breast cancer-related lymphedema and quality of life: A randomized controlled trial. Eur J Oncol Nurs. 2019 Jun;40:22-35. doi: 10.1016/j.ejon.2019.02.006. Epub 2019 Feb 25. PMID 31229204